CLINICAL TRIAL: NCT07287189
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Dose Comparison and Exploratory Efficacy Study of Orally Administered SAT-3247 in Ambulatory DMD Patients
Brief Title: Phase 2 Study of SAT-3247 in Pediatric Ambulatory Patients
Acronym: BASECAMP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Satellos Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAT-3247-CL-201; 2025-522522-13-01 (EU CTIS Number)
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy; Duchenne; DMD; Neuromuscular Diseases; Muscular Dystrophies
Keywords: muscle regeneration; satellite cell; asymmetric division; dystrophin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Neuromuscular Diseases; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, 2-dose comparison
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAT-3247 60 mg (Active Comparator): SAT-3247 60 mg oral tablets administered daily for 12 weeks
  Interventions: Drug: SAT-3247
- SAT-3247 120 mg (Active Comparator): SAT-3247 120 mg oral tablets administered daily for 12 weeks; note the 120 mg dose will not be studied in the US and Canada
  Interventions: Drug: SAT-3247
- placebo (Placebo Comparator): placebo oral tablets administered daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAT-3247 — SAT-3247 is a selective AAK1 inhibitor for oral tablet administration which promotes functional rescue of asymmetric satellite cell division, resulting in the robust production of muscle progenitor cells, subsequent improvement in muscle regeneration, and enhanced muscle function.
  Arms: SAT-3247 120 mg; SAT-3247 60 mg
Drug: Placebo — matching placebo oral tablets
  Arms: placebo

SUMMARY:
Phase 2a trial of SAT-3247 in ambulatory DMD patients aged ≥ 7 and < 10 years. The trial will study two doses of SAT-3247 in a randomized, double-blind, placebo-controlled weekday regimen for 12 weeks to determine the optimal dose, safety, tolerability, and preliminary efficacy.

DETAILED DESCRIPTION:
This is a global phase 2a trial of SAT-3247 in ambulatory DMD patients aged ≥ 7 and < 10 years. The trial will study two doses of SAT-3247 in a randomized, double-blind, placebo-controlled weekday regimen for 12 weeks to determine the optimal dose, safety, tolerability, and preliminary efficacy. One dose of SAT-3247 and placebo will be studied in the US and Canada; two doses of SAT-3247 and placebo will be studied in UK, EU, Serbia, and Australia.

Enrollment of up to 51 ambulatory DMD participants aged ≥ 7 and < 10 years of age is planned globally. Randomization will be stratified by baseline corticosteroid regimen and prior DMD concomitant medications.

Each participant will receive once daily doses of SAT-3247 or matched placebo for 12 weeks.

Participants will be screened within 28 days before initiating dosing of investigational product at Baseline. Following the Screening period, participants will complete a Baseline visit (Visit 2), a follow-up phone call at Week 1, and visits at Week 4 (Visit 3), Week 8 (Visit 4), and Week 12 (Visit 5).

ELIGIBILITY:
Key Inclusion Criteria:

* Has a definitive diagnosis of DMD based on documented clinical findings and prior genetic testing with a confirmed mutation in the DMD gene.
* Male DMD patients who are ambulatory and aged ≥ 7 to < 10 years at the time of screening.
* Stable dose of systemic glucocorticoids (i.e., prednisolone, deflazacort, or vamorolone) according to the standard of care for ≥ 3 months prior to the Screening Visit and for the duration of the trial. Patients who are not receiving glucocorticosteroids are also eligible if stopped ≥ 3 months prior to the Screening Visit.
* Stable doses of prescription medicines including ACE inhibitors, β-blockers, and diuretics (excluding glucocorticosteroids) and over-the-counter medicines and/or herbal supplements for supportive care ≥ 1 month prior to the Screening Visit and for the duration of the trial.
* Participants that have previously received delandistrogene moxeparvovec (brand name Elevidys) either in a prior clinical trial or in the commercial setting > 18 months prior to screening whose muscle function tests have stabilized or demonstrated decline ≥ 3 months prior to Screening, as determined by investigator and documented in chart notes, will be eligible.
* Participants that have previously received an exon skipper > 6 months prior to Screening whose muscle function tests have stabilized or demonstrated decline ≥ 3 months prior to Screening, as determined by investigator and documented in chart notes, will be eligible.
* Participants receiving a stable dose of givinostat (brand name Duvyzat) for at least 18 months or longer prior to the Screening Visit will be eligible. Participants unable to tolerate givinostat who discontinued treatment before 18 months are eligible to enroll if date of last dose is ≥ 30 days from the Screening date. Givinostat should not be discontinued, if tolerated, to meet study entry criteria.
* Participants that have received prior treatment with an investigational gene therapy product (other than delandistrogene moxeparvovec) ≥ 24 months prior to the Screening Visit.
* If participating in a physical therapy/strength training regimen, must be stable for ≥ 2 months prior to the Screening Visit and for the duration of the trial.

Key Exclusion Criteria:

* Ambulatory patients expected to experience loss of ambulation within ≤ 12 months.
* Participants for whom MRI or open muscle biopsy are contraindicated.
* Evidence of significant hepatic dysfunction, defined as GLDH > 2X upper limit of normal (ULN) at the Screening Visit.
* Impaired cardiac function defined as a left ventricular ejection fraction of < 50% on screening cardiac assessments (echocardiogram or MRI) or evidence of symptomatic cardiomyopathy.
* A forced vital capacity < 60% predicted at the Screening Visit.
* Ongoing participation in any other therapeutic clinical trial or follow-up study for a therapeutic intervention
* Consumption of grapefruit juice or grapefruit containing products
* Severe behavioural or cognitive problems that preclude participation in the study, in the opinion of the investigator.

Additional entry criteria will be reviewed with the clinical site investigator.

Ages: 7 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — gender assigned at birth
Enrollment: 51 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of SAT-3247 | 12 weeks
  Occurrence of treatment emergent adverse events and relationship to investigational product
Tolerability of SAT-3247 | 12 weeks
  occurrence of clinically significant changes in physical exam, clinical laboratory measures, vital signs, and ECG
SAT-3247 effects on muscle strength | 12 weeks
  change from baseline in muscle force as determined by dynamometry

SECONDARY OUTCOMES:
SAT-3247 effects on muscle quality | 12 weeks
  change from baseline in intramuscular fat fraction in quantitative magnetic resonance in vastus lateralis (thigh muscle)
SAT-3247 effects on muscle function | 12 weeks
  changes from baseline in north star ambulatory assessment
SAT-3247 effects on muscle function | 12 weeks
  changes from baseline in stride velocity 95th Centile
SAT-3247 effects on muscle regeneration | 12 weeks
  changes from baseline in the regeneration index as measured from an open biopsy of biceps brachii

CONTACTS AND LOCATIONS:
Overall Officials: Satellos Chief Medical Officer, Study Director — Satellos Bioscience, Inc.
Locations (18):
- United States (11):
  - University of California Los Angeles, Los Angeles, California
  - Colorado Children's, Aurora, Colorado
  - Lurie Children's, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Washington University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's, Seattle, Washington
- Australia (2):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital Melbourne, Melbourne, Victoria
- Children's Hospital Eastern Ontario, Ottawa, Ontario, Canada
- Serbia (3):
  - Clinic of Neurology and Psychiatry for Children and Youth, Belgrade
  - University Children's Clinic Tirsova, Belgrade
  - Mother and Child Health Care Institute, Belgrade
- Great Ormond Street, London, UK, United Kingdom